CLINICAL TRIAL: NCT07349576
Title: Precision Dietary Intervention Improves Postoperative Energy Intake, Nutritional Status, and Recovery in Patients Undergoing Hepatectomy for Liver Cancer: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Provincial Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024KY-013
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Primary Liver Cancer
Keywords: Primary liver cancer;Hepatectomy;Precision diet;Early feeding;Postoperative rehabilitation;Nutritional care
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dietary intervention group (Experimental)
  Interventions: Dietary Supplement: Special diet plan and whole protein preparation NUTRICIA for 5 days after liver resection for liver cancer
- standard care group (Experimental)
  Interventions: Other: Conventional dietary intervention

INTERVENTIONS:
Dietary Supplement: Special diet plan and whole protein preparation NUTRICIA for 5 days after liver resection for liver cancer — The intervention group, based on the control group, followed the "Chinese Clinical Practice Guidelines for Enhanced Recovery After Surgery (Part II)"and evidence-based summaries, combined with the "Chinese Expert Consensus on Perioperative Management for Hepatectomy in Hepatocellular Carcinoma (2021 Edition)" and oral nutritional supplementation guidelines, Based on the patient's comorbidities, liver characteristics, and gastrointestinal recovery patterns, a specialized 5-day post-hepatectomy diet plan for liver cancer patients has been developed. Postoperatively, oral nutritional supplements (ONS) were administered at 9:30 AM and 3:00 PM between meals, and at 9:00 PM after dinner, using the whole protein preparation NUTRICIA(specification: 320g/can, manufacturer: Milupa GmbH, Germany, production batch: HJ20170172).
  Arms: dietary intervention group
Other: Conventional dietary intervention — After returning to the ward after the operation under the traditional dietary guidance model, the patient regained consciousness under anesthesia without nausea, vomiting, etc., and began to try drinking water. If there are no special conditions such as gastrointestinal discomfort, then starting according to the dietary principles, that is, a liquid diet on the first day after the operation, a semi-liquid diet on the second day, and gradually transitioning to a regular diet from the third day after the operation until discharge based on the patient's tolerance. One to two days after the operation, parenteral nutrition mixtures are routinely infused.
  Arms: standard care group

SUMMARY:
Objective:To explore the application effect of postoperative refined early dietary plan in the enhanced recovery of patients undergoing hepatectomy for primary liver cancer, and to provide scientific evidence for optimizing postoperative dietary structure and increasing oral energy intake of patients.

Methods:In this randomized, parallel-controlled trial, 142 colorectal cancer survivors meeting inclusion criteria were recruited from a tertiary hospital in Hefei, Anhui Province. Participants were randomly assigned in a 1:1 ratio to either the dietary intervention group or the conventional diet group. Both the standard care group and the dietary intervention group received 5 days of routine dietary care. The dietary intervention group additionally received specialized meal plans and whole protein supplements beyond the standard care regimen. Dietary intake, nutritional status, and postoperative recovery outcomes were measured and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* (1) Pathologically confirmed diagnosis of primary hepatocellular carcinoma; (2) Underwent elective (partial) hepatectomy; (3) Age 18-80 years; (4) Basically normal renal function and preoperative Child-Pugh liver function grade A or B; (5) Voluntary participation in the study and signed informed consent.

Exclusion Criteria:

* (1) Concurrent malignant tumors; (2) Postoperative deterioration or contraindications to oral intake (e.g., dysphagia, intestinal obstruction); (3) Severe malnutrition or other disorders affecting nutritional metabolism; (4) Major intraoperative complications (e.g., massive hemorrhage, bile leakage, intra-abdominal adhesions); (5) Postoperative transfer to the ICU.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2024-01-04 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Prealbumin | Six days after the operation
albumin | Six days after the operation

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Provincal Hospital, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: Undecided